CLINICAL TRIAL: NCT06358118
Title: Clinical Research on Evidence Based Traditional Chinese Medicine for Elderly Diabetes Based on State Target Theory-Buyuan Zhixiao Fang in the Treatment of Elderly Patients With Diabetes and Multiple Metabolic Disorders: Study Protocol for a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Buyuan-zhixiao Formula in the Treatment of Elderly Patients With Diabetes and Multiple Metabolic Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qing Ni (Other)
Responsible Party: Sponsor-Investigator, Qing Ni, Clinical Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-003-KY
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Diabete Mellitus; Aging; Metabolic Disorders; Traditional Chinese Medicine; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Take Buyuan Zhixiao Formula granules
  Interventions: Drug: Buyuan Zhixiao Formula
- control group (Placebo Comparator): Take a placebos
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buyuan Zhixiao Formula — Buyuan Zhixiao Formula
  Arms: experimental group
Drug: Placebo — The placebo contains 10% of the active ingredients of the Chinese medicine group
  Arms: control group

SUMMARY:
The primary objective of this clinical trial is to assess the clinical efficacy and safety of the Buyuan Zhixiao Formula in treating elderly patients with diabetes and multiple metabolic disorders exhibiting symptoms of renal deficiency and blood stasis. Furthermore, this study aims to intervene in high-risk factors to prevent arteriosclerosis and to investigate the clinical efficacy of the Buyuan Zhixiao Formula in the prevention and treatment of cognitive impairments.

The main questions it aims to answer are:

1. What are the clinical effects of Buyuan Zhixiao Formula, including lowering blood sugar, lowering blood pressure, lowering lipids, and treating obesity?
2. Can Buyuan Zhixiao Formula improve cognitive impairment in diabetes? Researchers compared Buyuan Zhixiao Formula with a placebo (a drug that looks similar but contains only 10% of the active ingredients) to see if the drug Buyuan Zhixiao Formula can treat elderly people with diabetes and multiple metabolic disorders.

Participants will:

1. Take the drug Bu Yuan Zhi XiaoFormula or placebo every day for 6 months；Follow-up for 6 months；
2. Check fasting blood sugar and 2-hour postprandial blood sugar every month; check HbA1c, blood lipids, vascular function, and cognitive impairment serum markers every 3 months;
3. Conduct scores on TCM symptoms, cognitive ability, nutritional status and other scales and adverse events;
4. Urine and serum samples were collected before and after treatment;

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥65 years, irrespective of sex;
* 2.Individuals who meet the Western medical diagnostic criteria for type 2 diabetes mellitus (T2DM) in the elderly, with a hemoglobin A1c level of ≥7.0% in the past three months;
* 3.Compliance with the diagnostic criteria for abdominal obesity (waist circumference ≥90 cm for males and ≥85 cm for females);
* 4.Conformity to the diagnostic standards for hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg);
* 5.A history of dyslipidemia, where lipid levels have not reached the general control standards for elderly individuals with T2DM following oral lipid-lowering therapy (statins/bile acid sequestrants): LDL cholesterol <2.6 mmol/L and/or triglycerides <2.5 mmol/L;
* 6.Diagnosis of kidney deficiency and blood stasis according to traditional Chinese medicine, with the pattern type referring to the《Guidelines for Clinical Research of New Chinese Medicines》;
* 7.Willingness to sign an informed consent document.

Exclusion Criteria:

* 1.Exclusion of individuals who, within the past week, have experienced severe infections, acute cardiovascular or cerebrovascular events (such as acute cerebral infarction or myocardial infarction), significant trauma, acute pancreatitis, or other conditions that could precipitate stress-induced hyperglycemia. This also extends to those with concurrent endocrinopathies that may induce insulin resistance, such as Cushing's syndrome, hyperthyroidism, or pituitary growth hormone adenomas, as well as those currently receiving treatment with glucocorticoids or undergoing chemotherapy for malignancies.
* 2.Exclusion of individuals with a history of neurological disorders or psychiatric conditions that could impair cognitive function, as well as those with a history of medication use for these conditions.
* 3.Exclusion of individuals with severe complications of diabetes such as diabetic nephropathy in the uremic stage, or those with significant primary diseases of the cardiovascular, cerebrovascular, hepatic, renal, or hematopoietic systems, as well as individuals diagnosed with cancer.
* 4.Exclusion of individuals with communication barriers that could affect the assessment of cognitive function, including severe impairments in speech, vision, and hearing.
* 5.Individuals who have participated in other pharmacological clinical trials within the past month.
* 6.Individuals who have insufficient understanding of this study, are unwilling to participate, or, based on the researchers' judgment, present a reduced likelihood of enrollment or poor compliance due to unstable work and living locations or other factors that could lead to loss to follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-06 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Measured at 0, 3, 6, and 12 months respectively.
  unit：%

SECONDARY OUTCOMES:
Fasting blood glucose | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：mmol/l
2-hour postprandial blood glucose | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：mmol/l
blood pressure | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：mmHg
weight | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：KG
waist circumference | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：cm
BMI | Measured at 0, 1, 2, 3, 4, 5, 6, 9, and 12 months respectively
  unit：kg/m2
Total Cholesterol | Measured at 0, 3, 6, and 12 months
  unit：mmol/l
Triglycerides | Measured at 0, 3, 6, and 12 months
  unit：mmol/l
High density lipoprotein cholesterol | Measured at 0, 3, 6, and 12 months
  unit：mmol/l
Low density lipoprotein cholesterol | Measured at 0, 3, 6, and 12 months
  unit：mmol/l
Ankle-Brachial Index（ABI） | Measured at 0, 3, 6, and 12 months
  The normal range for the ABI is generally considered to be from 0.9 to 1.3.
Fasting insulin | Measured at 0, 3, 6, and 12 months
  unit：pmol/L
C-peptide | Measured at 0, 3, 6, and 12 months
  unit：pmol/L
insulin resistance index | Measured at 0, 3, 6, and 12 months
islet β-cell function index | Measured at 0, 3, 6, and 12 months
lipid Lipid accumulation product | Measured at 0, 3, 6, and 12 months
visceral adiposity index | Measured at 0, 3, 6, and 12 months
Measurement Results of Tumor Necrosis Factor-alpha Levels at Different Time Points | Measured at 0, 3, 6, and 12 months
Concentration Variation of Interleukin-10 | Measured at 0, 3, 6, and 12 months
Change in Homocysteine Levels | Measured at 0, 3, 6, and 12 months
Average Concentration of Interleukin-6 | Measured at 0, 3, 6, and 12 months
Change in Endothelin-1 Levels | Measured at 0, 3, 6, and 12 months
Average Concentration of Nitric Oxide | Measured at 0, 3, 6, and 12 months
Concentration Variation of Von Willebrand Factor | Measured at 0, 3, 6, and 12 months
Measurement Results of Vascular Endothelial Growth Factor Levels at Different Time Points | Measured at 0, 3, 6, and 12 months
Change in Matrix Metalloproteinase-9 Levels" or "Participants' Matrix Metalloproteinase-9 Concentration | Measured at 0, 3, 6, and 12 months
Average Concentration of Soluble Intercellular Adhesion Molecule-1 | Measured at 0, 3, 6, and 12 months
Change in Serum Tau Protein Levels | Measured at 0, 3, 6, and 12 months
Average Concentration of Aβ40 | Measured at 0, 3, 6, and 12 months
Average Concentration of Aβ42 | Measured at 0, 3, 6, and 12 months
Change in Neurofilament Light Chain Protein Levels | Measured at 0, 3, 6, and 12 months
Carotid Ultrasound; Carotid Intima-Media Thickness. | Measured at 0, 6, and 12 months
Activities of Daily Living Scale score; Fried Frailty Phenotype Scale; Mini Nutritional Rating Scale; MoCA scale score; Traditional Chinese Medicine Kidney Deficiency and Blood Stasis Syndrome Scale score. | Measured at 0, 3, 6, and 12 months
Montreal Cognitive Assessment Score | Measured at 0, 3, 6, and 12 months
  The maximum score is 30 points, and the higher the score, the better the cognitive function.
Fried Frailty Phenotype Scale | Measured at 0, 3, 6, and 12 months
  Those who have 5 or more of the items in the table can be diagnosed as frailty syndrome; those with less than 3 items are in the early stage of frailty; 0 items are healthy elderly people without frailty.
Activities of Daily Living Scale score | Measured at 0, 3, 6, and 12 months
  The scale consists of 10 items, with a total score of 100 points. The Cronbach's alpha of the scale is 0.813. A score of 100 points is considered normal, while scores below 100 indicate a decline.A score of 100 points indicates full independence in daily living, without any dependency; 61-99 points suggest mild dependency; 41-60 points indicate moderate dependency;
  ≤40 points denote severe dependency.
Mini Nutritional Rating Scale | Measured at 0, 3, 6, and 12 months
  The total score is 14 points, with the Cronbach's alpha of the scale being 0.906. A score of ≤7 points is considered malnourished, 8-11 points indicate a risk of malnutrition, and 12-14 points are indicative of normal nutrition.
  The total score is 14 points, with the Cronbach's alpha of the scale being 0.906. A score of ≤7 points is considered malnourished, 8-11 points indicate a risk of malnutrition, and 12-14 points are indicative of normal nutrition.
Serum and urine metabolomics | Measured at 0 and 6 months respectively
  Inferring the potential biological mechanisms of the effect of Buyuan Zhixiao Formula based on the differences in metabolic products in the blood and urine between the experimental and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Ni, postgraduate, Principal Investigator — China Academy of Chinese Medical Sciences Guang'anmen Hospital
Locations (6):
- China (6):
  - China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijin, Beijing Municipality
  - Cangzhou integrative medicine hospital, Hebei
  - Hohhot Mongolian Traditional Chinese Medicine Hospital, Neimeng
  - Binzhou Traditional Chinese Medicine Hospital, Shandong
  - Yantai Baishi Traditional Chinese Medicine Hospital, Shandong
  - The First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunes BP, Flores TR, Mielke GI, Thume E, Facchini LA. Multimorbidity and mortality in older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2016 Nov-Dec;67:130-8. doi: 10.1016/j.archger.2016.07.008. Epub 2016 Aug 2. PMID 27500661
- [Background] Quinones AR, Markwardt S, Botoseneanu A. Diabetes-Multimorbidity Combinations and Disability Among Middle-aged and Older Adults. J Gen Intern Med. 2019 Jun;34(6):944-951. doi: 10.1007/s11606-019-04896-w. Epub 2019 Feb 27. PMID 30815788
- [Background] Ji L, Hu D, Pan C, Weng J, Huo Y, Ma C, Mu Y, Hao C, Ji Q, Ran X, Su B, Zhuo H, Fox KA, Weber M, Zhang D; CCMR Advisory Board; CCMR-3B STUDY Investigators. Primacy of the 3B approach to control risk factors for cardiovascular disease in type 2 diabetes patients. Am J Med. 2013 Oct;126(10):925.e11-22. doi: 10.1016/j.amjmed.2013.02.035. Epub 2013 Jun 27. PMID 23810406
- [Background] Carnethon MR, Biggs ML, Barzilay J, Kuller LH, Mozaffarian D, Mukamal K, Smith NL, Siscovick D. Diabetes and coronary heart disease as risk factors for mortality in older adults. Am J Med. 2010 Jun;123(6):556.e1-9. doi: 10.1016/j.amjmed.2009.11.023. PMID 20569763
- [Background] Al Slail FY, Abid O, Assiri AM, Memish ZA, Ali MK. Cardiovascular risk profiles of adults with type-2 diabetes treated at urban hospitals in Riyadh, Saudi Arabia. J Epidemiol Glob Health. 2016 Mar;6(1):29-36. doi: 10.1016/j.jegh.2015.07.004. Epub 2015 Aug 6. PMID 26257035
- [Result] Sinclair A, Saeedi P, Kaundal A, Karuranga S, Malanda B, Williams R. Diabetes and global ageing among 65-99-year-old adults: Findings from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2020 Apr;162:108078. doi: 10.1016/j.diabres.2020.108078. Epub 2020 Feb 14. PMID 32068097
- [Result] Al-Maskari F, El-Sadig M, Nagelkerke N. Assessment of the direct medical costs of diabetes mellitus and its complications in the United Arab Emirates. BMC Public Health. 2010 Nov 8;10:679. doi: 10.1186/1471-2458-10-679. PMID 21059202
- [Result] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Result] Ramtahal R, Khan C, Maharaj-Khan K, Nallamothu S, Hinds A, Dhanoo A, Yeh HC, Hill-Briggs F, Lazo M. Prevalence of self-reported sleep duration and sleep habits in type 2 diabetes patients in South Trinidad. J Epidemiol Glob Health. 2015 Dec;5(4 Suppl 1):S35-43. doi: 10.1016/j.jegh.2015.05.003. Epub 2015 Jun 11. PMID 26073574